CLINICAL TRIAL: NCT06717568
Title: Assessment of Adolescent Idiopathic Scoliosis Based on 3D Imaging Technology Using a Depth Camera
Brief Title: 3D Depth Camera-Based Assessment of Adolescent Idiopathic ScoliosisUsing a Depth Camera
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-KL-215-01-3
Record Dates: First submitted 2024-11-30; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- participant: BHD Measurement: Each participant undergoes two measurements by two different assessors, with a 5-minute interval between each measurement. The average value is taken.
  ATR Measurement: The trunk rotation angle (ATR) is measured using a Scoliometer. Two assessors each perform two measurements, with a 5-minute interval between each, and the average value is taken.
  Cobb Angle Measurement: Two experienced spinal specialists independently measure the Cobb angle, with each performing two measurements. The average value is taken. If their measurements differ by 5° or more, a third senior physician is required to perform a review.
  Interventions: Diagnostic Test: no intervention

INTERVENTIONS:
Diagnostic Test: no intervention — This is a diagnostic test with no intervention.

SUMMARY:
Adolescent Idiopathic Scoliosis (AIS) is a common spinal deformity affecting adolescent health, and early diagnosis and accurate assessment are crucial for preventing disease progression. Traditional assessment indicators, such as the trunk rotation angle (ATR) and Cobb angle, rely on clinical examinations and X-ray imaging, which have certain limitations, including radiation exposure and insufficient sensitivity. The Back Height Difference (BHD), as a quantitative measure of the back surface morphology, may reflect the degree of trunk deformity caused by scoliosis.

The use of the Kinect v2 depth camera to capture three-dimensional point cloud data of the back provides a high-precision, radiation-free assessment method.

ELIGIBILITY:
Inclusion Criteria:

(1) Adolescents aged 10-18 years, diagnosed with adolescent idiopathic scoliosis (AIS) with a Cobb angle ≥10°; (2) No history of spinal surgery or other corrective treatments; (3) Able to undergo short-term inpatient treatment (5 days) and comply with study procedures.

Exclusion Criteria:

(1) Patients with congenital, neuromuscular, or other secondary scoliosis; (2) Presence of major comorbidities affecting spinal structure or muscle tone (e.g., spinal cord injury, muscular dystrophy); (3) Patients unable to complete standardized assessment procedures.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study focuses on adolescents aged 10-18 diagnosed with adolescent idiopathic scoliosis, defined by a Cobb angle of ≥10°.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Back height difference | Day 1 of Admission
  Using depth cameras to acquire back data, point cloud processing algorithms analyze the information. The height difference between the highest point on the convex side and the corresponding point on the concave side is measured, with three repetitions taken to calculate the average value.

SECONDARY OUTCOMES:
Angle of trunk rotation | Day 1 of Admission
  A scoliometer is used to measure the patient's angle of trunk rotation (ATR). Measurements are repeated three times, and the average value is taken.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen S, Liu C, Mou J, Liang J, Sun Y, Chen X, Yu B, Li J, Zhu H, Pan Y, Du H. Radiation-free 3D assessment of back height differences via three-dimensional depth sensing in adolescent idiopathic scoliosis: prospective, single-center, observational study. Eur Spine J. 2025 Jul 21. doi: 10.1007/s00586-025-09154-8. Online ahead of print. PMID 40689983